CLINICAL TRIAL: NCT04055519
Title: Clinical Performance Assessment of a Daily Wear Monthly Replacement Soft Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLY935-C007
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Refractive Errors
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LID017569, then Biofinity (Other): Lehfilcon A contact lenses worn first, followed by comfilcon A contact lenses, as randomized. Each product will be worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses will be removed nightly for cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Comfilcon A contact lenses; Device: Multi-purpose disinfection solution
- Biofinity, then LID017569 (Other): Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each product will be worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses will be removed nightly for cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Comfilcon A contact lenses; Device: Multi-purpose disinfection solution

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Investigational silicone hydrogel contact lenses
  Other Names: LID017569
Device: Comfilcon A contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Biofinity®
Device: Multi-purpose disinfection solution — Solution for cleaning, disinfecting, and reconditioning silicone hydrogel contact lenses
  Other Names: OPTI-FREE® RepleniSH®

SUMMARY:
The purpose of this study is to obtain on-eye performance data to inform contact lens product development.

DETAILED DESCRIPTION:
Subjects are expected to attend 5 scheduled visits. The expected duration of subject participation in the study is approximately 60 days, with approximately 30 days (± 2 days) per product.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Successful wear of spherical weekly/monthly soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
* Possess spectacles that provide a corrected visual acuity of 20/40 or better in both eyes.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria

* Any eye condition or disease or use of medication that contraindicates contact lens wear.
* Eye surgery, irregular cornea, eye injury as specified in the protocol.
* Routinely sleeps in contact lenses at least 1 night per week over the last 3 months prior to enrollment.
* Any use of topical ocular medications, artificial tear or rewetting drops that would require instillation during contact lens wear.
* Habitually wears Biofinity contact lenses.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (3):
- United States (3):
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 3 investigative sites located in the US.
Pre-assignment Details: This reporting group includes all randomized subjects/eyes (36/72) as treated. Note: Two subjects received investigational product misallocations and were exposed to the incorrect study product in the sequence.
Units Other Than Participants: eyes
Groups:
- LID017569, Then Biofinity: Lehfilcon A contact lenses worn in Period 1, with comfilcon A contact lenses worn in Period 2, as randomized. Each product was worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses were removed nightly for cleaning and disinfection.
- Biofinity, Then LID017569: Comfilcon A contact lenses worn in Period 1, with lehfilcon A contact lenses worn in Period 2, as randomized. Each product was worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses were removed nightly for cleaning and disinfection.
Period: First Wear Period (30 Days)
Arm/Group | LID017569, Then Biofinity | Biofinity, Then LID017569
Started | 16; 32 eyes | 20; 40 eyes
Completed | 16; 32 eyes | 20; 40 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Second Wear Period (30 Days)
Arm/Group | LID017569, Then Biofinity | Biofinity, Then LID017569
Started | 16; 32 eyes | 20; 40 eyes
Completed | 16; 32 eyes | 20; 40 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects exposed to any study lenses evaluated in this study.
Groups:
- Overall: LID017569 and Biofinity contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized. Each product was worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses were removed nightly for cleaning and disinfection.
Arm/Group | Overall
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Distance VA (logMAR) With Study Lenses
Description: Visual acuity (VA) was collected for each eye individually with study lenses in place at a distance of 4 meters using a letter chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Day 30 after a minimum of 6 hours of wear, each product
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID017569: Lehfilcon A contact lenses worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses were removed nightly for cleaning and disinfection.
- Biofinity: Comfilcon A contact lenses worn in both eyes on a daily wear basis at least 8 hours a day, 5 days a week, for 30 days. Lenses were removed nightly for cleaning and disinfection.
Arm/Group | LID017569 | Biofinity
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 72 | 72
logMAR | -0.13 (0.06) | -0.14 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 60 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes were categorized under the actual study lenses exposed in the corresponding lens sequence.
Groups:
- Pre-treatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID017569 Ocular; LID017569 Nonocular/Systemic: Events reported in this group occurred while exposed to lehfilcon A contact lenses
- Biofinity Ocular; Biofinity Nonocular/Systemic: Events reported in this group occurred while exposed to comfilcon A contact lenses
Arm/Group | Pre-treatment | LID017569 Ocular | LID017569 Nonocular/Systemic | Biofinity Ocular | Biofinity Nonocular/Systemic
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/72 | 0/36 | 0/72 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/72 | 0/36 | 0/72 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/72 | 0/36 | 0/72 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT04055519/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT04055519/SAP_001.pdf